CLINICAL TRIAL: NCT02879136
Title: TAME-PD - Physical Therapy, Atomoxetine and, Methylphenidate, to Enhance Gait and Balance in Parkinson's Disease: A Single Center, Randomized Pilot Study
Brief Title: TAME-PD - Physical Therapy, Atomoxetine and, Methylphenidate, to Enhance Gait and Balance in Parkinson's Disease
Acronym: TAME-PD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hubert Fernandez (Other)
Responsible Party: Sponsor-Investigator, Hubert Fernandez, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-277
Record Dates: First submitted 2016-06-23; First posted 2016-08-25 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease, Idiopathic
Keywords: Gait; Balance; PD
MeSH Terms: conditions — Parkinson Disease | interventions — Methylphenidate; Physical Therapy Modalities; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical Therapy (Active Comparator): Physical Therapy (PT) will consist of two weekly sessions over a 12 week period using the Mellen center protocol PT for PD.
  Interventions: Other: Physical Therapy
- Physical Therapy plus Methylphenidate (Active Comparator): Methylphenidate 20 mg daily in combination with PT
  Interventions: Drug: Methylphenidate; Other: Physical Therapy
- Physical Therapy plus Atomoxetine (Active Comparator): Atomoxetine 10 mg daily in combination with PT or PT alone.
  Interventions: Other: Physical Therapy; Drug: Atomoxetine

INTERVENTIONS:
Drug: Methylphenidate — Patient will be randomized to Methylphenidate
  Other Names: Ritalin
  Arms: Physical Therapy plus Methylphenidate
Other: Physical Therapy — All Patients will have standard of care PT used for PD patients
  Other Names: PT
Drug: Atomoxetine — Patient will be randomized to Atomoxetine
  Other Names: Straterra
  Arms: Physical Therapy plus Atomoxetine

SUMMARY:
Gait and balance problems are a significant source of disability in patients with Parkinson disease. Physical therapy remains one of the main treatments. On the other hand some medications, such as methyphenidate and atomoxetine, have been tried with promising results. The outcomes in gait and balance in Parkinson disease after a combination of physical therapy and the medications mentioned above have not been explored yet. The investigators want to evaluate whether the addition of medication, either low dose of methylphenidate or atomoxetine, to physical therapy will achieve improvement in gait and balance in Parkinson disease more than physical therapy alone. The investigators propose a pilot, single center, rater blind, prospective randomized trial. 2-arm-parallel group, intention-to-treat analysis.

DETAILED DESCRIPTION:
Gait impairment and postural instability constitute major sources of disability in Parkinson disease (PD). Increased level of dependence in activities of daily living and augmented risk of falling are the main consequences. About 87% of patients experience at least one fall during their illness, 65% an injury that requires evaluation in an emergency room, and up to 33% sustain one or more fractures.

Pedunculopontine nucleus, locus ceruleus, frontal brain cortex, and striatum play a critical role in gait and balance, with dopamine, noradrenaline and acetylcholine as the main neurotransmitters. Therefore, increased availability of dopamine in the nigrostriatal pathway, and enhanced disposal of central noradrenaline and acetylcholine in the locus ceruleus can in theory, contribute to improvement .

Methylphenidate and atomoxetine are dopamine and noradrenaline reuptake inhibitors approved for the treatment of attention disorders. Interestingly, growing literature suggests a promising role of these medications in gait and balance in PD. Three open-label studies reported efficacy of methylphenidate in gait impairment in patients with PD. Auriel et al used a single 20 mg dose of methylphenidate in 23 patients and found an improvement in gait speed, stride time variability, and timed gait. In a second study, 5 patients received a single 10-mg dose of methylphenidate and improvements were noted in total walking time, total freezing time, number of freezing episodes, and nonfreezing walking time. Another study, which evaluated a 50 to 80 mg dose of methylphenidate over 3 months in 17 patients undergoing concomitant deep brain stimulation, found an improvement in both timed gait and in the number of freezing episodes.

However, the only randomized clinical trial with methylphenidate showed a different result. Twenty-three subjects with PD and moderate gait impairment were screened for this 6- month, placebo-controlled, double-blind study. Subjects were randomly assigned to high dose of methylphenidate (maximum, up to 80 mg/day) or placebo for 12 weeks and crossed over after a 3-week washout. The primary outcome measure was change in a gait composite score obtained through GAITrite (a system that was developed to measure and record temporal and spatial parameters of gait by using a walkway approximately 3 meters long with grids of embedded, pressure-sensitive sensors connected to a personal computer). Seventeen patients completed the trial. There was no change in the gait composite score or any of the secondary or exploratory variables such as fatigue, freezing, depression and daily sleepiness at 12 weeks; however, some improvement was noted in the early phase of the study.

The discrepancy between the results of the open label studies and the randomized study may be explained by dose of methylphenidate substantially higher in the RCT compared to the first two open-label studies. Whereas patients in the RCT received at least 65 mg/day, patients in the first two open-label studies received 10-20 mg/day. It is been suggested that the efficacy of methylphenidate and atomoxetine varies according to the dose administrated. The complex pharmacodynamic of dopamine and noradrenaline reuptake inhibitors in the presence of other dopaminergic therapies such as Levodopa or dopamine agonist, can elicit differences in response regarding the administered dose . During the early phase of the RCT when a trend improvement was noted, smaller doses of methylphenidate were being used as the patients were being titrated to their final dose. Low chronic doses of methylphenidate have not been tested to improve gait and balance in PD in any trial.

In the one pilot study thus far evaluating atomoxetine for gait freezing, a trend towards improvement in the gait and balance scale (GABS) was noted. However, this study was underpowered as only five patients participated in the study .

Simultaneously, diverse modalities of physical therapy (PT) have shown improvement in gait and balance in PD. A systematic review from Cochrane database concluded that different physiotherapy interventions were better than placebo over three months, in terms of velocity, two- or six-minute walk test, step length, Timed Up & Go, Functional Reach Test, Berg Balance Scale and clinician-rated UPDRS. The grade of improvement varied depending on the intervention and outcome measure, ranging from 10 to 30%.

To the best of the investigators' knowledge, the combination of medication and physical therapy has never been evaluated previously in gait and balance in PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD having significant balance or gait disorder with a score ≥2 in the Unified Parkinson Disease Rating Scale (UPDRS) 3.10 item 'independent walking but with substantial gait impairment; not related to off periods' occurring despite satisfactory motor control by dopaminergic therapy, with a medication regimen unlikely to change in the next 30 days.

Exclusion Criteria:

* Previous participation in PD-specific PT.
* Presence of signs and symptoms suggestive of atypical parkinsonism.
* Concomitant conditions that may affect significantly the evaluation of balance or gait, including orthopedic, rheumatologic or other neurological diseases.
* Contraindication for physical therapy
* Comorbidities that contraindicate the use of the methylphenidate or atomoxetine: history of substance abuse, current severe anxiety, depression or psychosis, epilepsy, hyperthyroidism, glaucoma, cardiac arrhythmia, history of Tourette syndrome, hepatic disease, allergy to methylphenidate or atomoxetine.
* Concurrent use of MAO inhibitors, or use in the last two weeks.
* Previous deep brain stimulation procedure.
* Punctuation of 5 in Hoehn and Yard modified scale: 'Wheelchair bound or bedridden unless aided'.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation | 12 weeks
  Change in the balance evaluation systems test, MiniBest is standard gait analysis measure conducted by physical therapists.

SECONDARY OUTCOMES:
Change in gait | 12 weeks
  Stride length and gait velocity measured using "GaitRite", which is a standard gait analysis measure conducted by physical therapists.

OTHER OUTCOMES:
Motor function | 12 weeks
  UPDRS part III scale

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Fernandez, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boonstra TA, van der Kooij H, Munneke M, Bloem BR. Gait disorders and balance disturbances in Parkinson's disease: clinical update and pathophysiology. Curr Opin Neurol. 2008 Aug;21(4):461-71. doi: 10.1097/WCO.0b013e328305bdaf. PMID 18607208
- [Background] Williams DR, Watt HC, Lees AJ. Predictors of falls and fractures in bradykinetic rigid syndromes: a retrospective study. J Neurol Neurosurg Psychiatry. 2006 Apr;77(4):468-73. doi: 10.1136/jnnp.2005.074070. PMID 16543524
- [Background] Moreau C, Cantiniaux S, Delval A, Defebvre L, Azulay JP. [Gait disorders in Parkinson's disease: and pathophysiological approaches]. Rev Neurol (Paris). 2010 Feb;166(2):158-67. doi: 10.1016/j.neurol.2009.05.010. Epub 2009 Jul 18. French. PMID 19616816
- [Background] Wielinski CL, Erickson-Davis C, Wichmann R, Walde-Douglas M, Parashos SA. Falls and injuries resulting from falls among patients with Parkinson's disease and other parkinsonian syndromes. Mov Disord. 2005 Apr;20(4):410-415. doi: 10.1002/mds.20347. PMID 15580552
- [Background] Collomb-Clerc A, Welter ML. Effects of deep brain stimulation on balance and gait in patients with Parkinson's disease: A systematic neurophysiological review. Neurophysiol Clin. 2015 Nov;45(4-5):371-88. doi: 10.1016/j.neucli.2015.07.001. Epub 2015 Aug 28. PMID 26319759
- [Background] Nutt JG, Horak FB, Bloem BR. Milestones in gait, balance, and falling. Mov Disord. 2011 May;26(6):1166-74. doi: 10.1002/mds.23588. PMID 21626560
- [Background] Auriel E, Hausdorff JM, Herman T, Simon ES, Giladi N. Effects of methylphenidate on cognitive function and gait in patients with Parkinson's disease: a pilot study. Clin Neuropharmacol. 2006 Jan-Feb;29(1):15-7. doi: 10.1097/00002826-200601000-00005. PMID 16518128
- [Background] Pollak L, Dobronevsky Y, Prohorov T, Bahunker S, Rabey JM. Low dose methylphenidate improves freezing in advanced Parkinson's disease during off-state. J Neural Transm Suppl. 2007;(72):145-8. doi: 10.1007/978-3-211-73574-9_17. PMID 17982887
- [Background] Devos D, Krystkowiak P, Clement F, Dujardin K, Cottencin O, Waucquier N, Ajebbar K, Thielemans B, Kroumova M, Duhamel A, Destee A, Bordet R, Defebvre L. Improvement of gait by chronic, high doses of methylphenidate in patients with advanced Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 May;78(5):470-5. doi: 10.1136/jnnp.2006.100016. Epub 2006 Nov 10. PMID 17098845
- [Background] Espay AJ, Dwivedi AK, Payne M, Gaines L, Vaughan JE, Maddux BN, Slevin JT, Gartner M, Sahay A, Revilla FJ, Duker AP, Shukla R. Methylphenidate for gait impairment in Parkinson disease: a randomized clinical trial. Neurology. 2011 Apr 5;76(14):1256-62. doi: 10.1212/WNL.0b013e3182143537. PMID 21464430
- [Background] Mendonca DA, Menezes K, Jog MS. Methylphenidate improves fatigue scores in Parkinson disease: a randomized controlled trial. Mov Disord. 2007 Oct 31;22(14):2070-6. doi: 10.1002/mds.21656. PMID 17674415
- [Background] Jankovic J. Atomoxetine for freezing of gait in Parkinson disease. J Neurol Sci. 2009 Sep 15;284(1-2):177-8. doi: 10.1016/j.jns.2009.03.022. Epub 2009 Apr 9. PMID 19361809
- [Background] Mirelman A, Maidan I, Deutsch JE. Virtual reality and motor imagery: promising tools for assessment and therapy in Parkinson's disease. Mov Disord. 2013 Sep 15;28(11):1597-608. doi: 10.1002/mds.25670. PMID 24132848
- [Background] Gisbert R, Schenkman M. Physical therapist interventions for Parkinson disease. Phys Ther. 2015 Mar;95(3):299-305. doi: 10.2522/ptj.20130334. Epub 2014 Nov 25. No abstract available. PMID 25425695
- [Background] Tomlinson CL, Patel S, Meek C, Clarke CE, Stowe R, Shah L, Sackley CM, Deane KH, Herd CP, Wheatley K, Ives N. Physiotherapy versus placebo or no intervention in Parkinson's disease. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD002817. doi: 10.1002/14651858.CD002817.pub2. PMID 22786482
- [Background] Thomas M, Jankovic J, Suteerawattananon M, Wankadia S, Caroline KS, Vuong KD, Protas E. Clinical gait and balance scale (GABS): validation and utilization. J Neurol Sci. 2004 Jan 15;217(1):89-99. doi: 10.1016/j.jns.2003.09.005. PMID 14675615
- [Background] Williams JR, Hirsch ES, Anderson K, Bush AL, Goldstein SR, Grill S, Lehmann S, Little JT, Margolis RL, Palanci J, Pontone G, Weiss H, Rabins P, Marsh L. A comparison of nine scales to detect depression in Parkinson disease: which scale to use? Neurology. 2012 Mar 27;78(13):998-1006. doi: 10.1212/WNL.0b013e31824d587f. Epub 2012 Mar 14. PMID 22422897
- [Background] Leentjens AF, Dujardin K, Pontone GM, Starkstein SE, Weintraub D, Martinez-Martin P. The Parkinson Anxiety Scale (PAS): development and validation of a new anxiety scale. Mov Disord. 2014 Jul;29(8):1035-43. doi: 10.1002/mds.25919. Epub 2014 May 23. PMID 24862344